CLINICAL TRIAL: NCT01332448
Title: Meta-analysis of Orlistat Laboratory Data From Placebo-controlled Clinical Trials
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114237
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Obesity
Keywords: Xenical; Alli; safety; meta-analysis; liver-function test; Roche; orlistat
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Orlistat 120: Orlistat 120mg tid
  Interventions: Drug: Orlistat 120
- Orlistat 60: Orlistat 60 mg tid
  Interventions: Drug: Orlistat 60
- Placebo: No active drug
  Interventions: Drug: Orlistat 120; Drug: Orlistat 60

INTERVENTIONS:
Drug: Orlistat 120 — Orlistat 120mg tid
  Groups: Orlistat 120; Placebo
Drug: Orlistat 60 — Orlistat 60mg tid
  Groups: Orlistat 60; Placebo

SUMMARY:
Roche and GSK will carry out a meta-analysis of liver function data from trials of orlistat to establish whether there is any indication of liver toxicity. The motivation is a cumulative assessment of drug-induced liver injury (DILI) conducted by the FDA following spontaneous reports of liver toxicity in people taking Xenical or Alli.

ELIGIBILITY:
Inclusion Criteria:

1. The trial must be randomized and placebo-controlled
2. The orlistat dose must be 60mg or 120mg
3. Data on ALT or BIL must be available
4. The nominal treatment period must be 16 weeks or longer

Exclusion Criteria:

1. If cross-over trials are found, data from other than the first period will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All clinical trials found by search procedure:
  1. In-house trial repositories at GSK and Roche
  2. EMBASE (which includes MEDLINE) using the terms "orlistat", "Xenical" or "Alli", with "placebo" and "clinical trial"
  3. Recently published meta-analyses found by the search will also be searched for relevant trials
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Odds ratio (Orlistat120:Placebo) for subjects experiencing alanine transaminase (ALT) greater than upper limit of normal (ULN) | within one year of starting treatment
Odds ratio (Orlistat120:Placebo) for subjects experiencing total bilirubin (BIL) > ULN | within one year of starting treatment
Odds ratio (Orlistat120:Placebo) for subjects experiencing ALT > ULN for successive measurements more than two weeks apart | within one year of starting treatment
Odds ratio (Orlistat120:Placebo) for subjects experiencing BIL > ULN for successive measurements greater than two weeks apart | within one year of starting treatment

SECONDARY OUTCOMES:
Odds ratio (Orlistat60:Placebo) for subjects experiencing ALT > ULN | within one year of starting treatment
Odds ratio (Orlistat60:Placebo) for subjects experiencing BIL > ULN | within one year of starting treatment
Odds ratio (Orlistat60:Placebo) for subjects experiencing ALT > ULN for successive measurements more than two weeks apart | within one year of starting treatment
Odds ratio (Orlistat60:Placebo) for subjects experiencing BIL > ULN for successive measurements greater than two weeks apart | within one year of starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline